CLINICAL TRIAL: NCT04225689
Title: The Intensive Post Exclusive Enteral Nutrition Study (iPENS): A Randomised Trial to Evaluate CD-TREAT Diet as a Food Reintroduction Regime in Children and Young Adults With Crohn's Disease
Brief Title: The Intensive Post Exclusive Enteral Nutrition Study
Acronym: iPENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GN19GA433P
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Crohn Disease
Keywords: food reintroduction; dietary intervention; dietary triggers; faecal calprotectin; CD-TREAT; Exclusive enteral nutrition
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Masking Description: Electronic random block-size randomisation will be performed by a researcher not involved in study recruitment. Allocation to study arm will be revealed to participants after provision of informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD-TREAT diet (Experimental): Solid food-based dietary intervention replicating composition of exclusive enteral nutrition (EEN).
  Daily for a maximum of 21 days. Individualised diet based on energy requirements and physical activity levels.
  Interventions: Other: CD-TREAT diet
- Unrestricted diet (No Intervention): Free, unrestricted diet. Daily for a maximum of 21 days.

INTERVENTIONS:
Other: CD-TREAT diet — Dietary intervention
  Arms: CD-TREAT diet

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory condition with phases where the disease is active and other, where there are no symptoms. Exclusive enteral nutrition (EEN), a liquid only diet without allowance of any extra food, is the main treatment for children with active CD. However, when children stop the liquid diet and return to their normal diet, most of them will experience an increase in their gut inflammation, mostly without symptoms initially. The aim of this study is to investigate this phenomenon by exploring if diet and gut bacteria play a role. Furthermore, the investigators aim to test whether a new, ordinary food-based diet, called the Crohn's Disease TReatment with EATing (CD-TREAT) diet can help control gut inflammation during the early food reintroduction phase, after EEN completion, compared to an unrestricted, free diet.

DETAILED DESCRIPTION:
A maximum of 60 participants, who have successfully responded to EEN, will be allocated to the study arms with block randomisation, with a 1:1 allocation, in random size blocks. The electronic randomisation process will be performed by an independent researcher. Those participants who do not wish to be randomised to one of the two study arms, will be offered the chance to be allocated to the group of their preference. Using this approach, inclusion of all eligible participants will be ensured, as excluding those who do not wish to be randomised, may reduce the generalisation of findings and minimise statistical power of a study with modest eligible population to recruit from.

CD-TREAT diet (intervention group)

Participants in the intervention group will consume the CD-TREAT diet exclusively without being allowed to consume additional food, for the first 3 weeks of food reintroduction, after EEN completion. They will be provided with a tailored, dietitian-devised diet, which has been designed to replicate the nutritional composition of EEN. The intervention will be overseen by qualified dietitians, including a National Health Service (NHS) research dietitian.

Unrestricted diet (control group)

Participants in the control group will consume a free, unrestricted diet for the same period, as the intervention group.

Participants in both groups will record their diet on a daily basis. The investigators will meet the participants weekly to address any potential issues they may have during the trial and to review the dietary assessment process. Standard treatment for maintenance of clinical remission will be continued, as designated by the medical team.

Participants will be asked to provide serial faecal and urine samples (n=8). Collection of a maximum of 2 blood samples, anthropometric measurements and assessment of disease activity and quality of life will be performed before and after the end of the dietary intervention. Participants will also be followed through their clinical records until they clinically relapse, or maximum up to a year after EEN completion.

The primary endpoint is the comparison of faecal calprotectin levels between the two groups at the end of the dietary intervention (3 weeks after EEN completion).

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed or relapsing patients with active CD, who have shown clinical improvement by the 4th week of EEN treatment

Exclusion Criteria:

1. Administration of another induction treatment (e.g. corticosteroids, biologic agents).
2. Lack of clinical improvement with EEN treatment, as assessed by the clinical team.
3. Enrolment in other studies investigating the efficacy of novel therapies for maintenance or induction of remission.
4. Patients or families unable to provide written consent for participation in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Colonic inflammation | Baseline to 21 days post EEN completion
  Comparison of faecal calprotectin levels between the intervention (CD-TREAT) and the control (unrestricted diet) group

SECONDARY OUTCOMES:
Diet and faecal microbiome | Baseline to 21 days post EEN completion
  Association of fermentable carbohydrates intake with relative abundance of faecal bacteria
Diet and faecal metabolome | Baseline to 21 days post EEN completion
  Association of fermentable carbohydrates intake with concentration of short chain fatty acids in stool
Crohn's Disease activity score | Baseline to 21 days post EEN completion
  Comparison of weighted Paediatric Crohn's Disease Activity Index score between the two groups (minimum score: 0, maximum: 125). Higher score indicates higher disease activity severity.
Blood inflammatory markers | Baseline to 21 days post EEN completion
  Comparison of concentration of blood inflammatory cytokines between the two groups
Quality of life | Baseline to 21 days post EEN completion
  Comparison of IMPACT III scores between the two groups (minimum score: 35, maximum: 135). Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Russell, MBChB, MRCP, MRCPCH, PhD, Principal Investigator — NHS Greater Glasgow and Clyde; Konstantinos Gerasimidis, PhD, MSc, BSc, FHEA, Principal Investigator — University of Glasgow
Locations (5):
- United Kingdom (5):
  - University Hospital Crosshouse, Crosshouse
  - Royal Hospital for Sick Children, Edinburgh
  - Royal Hospital for Children, Glasgow
  - Forth Valley Royal Hospital, Larbert
  - University Hospital Wishaw, Wishaw

IPD SHARING:
Plan to Share IPD: Yes
Participants will be asked to provide written consent for their anonymised data to be made available to public data repositories.